CLINICAL TRIAL: NCT01685502
Title: Special Drug Use Investigation of Glucobay OD
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16517; Glucobay OD (Other: company internal)
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus
Keywords: Glucobay OD; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Acarbose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients treated with Glucobay OD under practical manner
  Interventions: Drug: Glucobay ODT (Acarbose, BAYG5421)

INTERVENTIONS:
Drug: Glucobay ODT (Acarbose, BAYG5421) — Patients treated with Glucobay OD under practical manner

SUMMARY:
The objective of this study is to assess the efficacy and safety under practical use of Glucobay OD. A total of 5,000 patients are to be enrolled to the study and assessed during 1 year observation period.

ELIGIBILITY:
Inclusion Criteria:

* Glucobay OD naive diabetics. patients with at least one of the following conditions: Uncontrollable with dietary therapy,exercise cure, diabetes medication, insulin therapy.

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Glucobay OD naive diabetics. Patients with at least one of the following conditions: Uncontrollable with dietary therapy,exercise cure, diabetes medication, insulin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2289 (Actual)
Dates: Start 2010-11; Primary Completion 2013-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) and serious adverse events (SAEs) | Up to 1 year
Decrease rate of HbA1c | Up to 1 year

SECONDARY OUTCOMES:
Body weight | up to1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan